CLINICAL TRIAL: NCT01390493
Title: Therapeutic Effects of Alpha-neurofeedback in the Treatment of Anorexia Nervosa
Brief Title: Therapeutic Effects of Neurofeedback in Anorexia Nervosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEUROAN
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Anorexia Nervosa
Keywords: neurofeedback, alpha, anorexia nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neurofeedback, alpha power (Experimental)
  Interventions: Behavioral: neurofeedback training

INTERVENTIONS:
Behavioral: neurofeedback training — training of individual alpha frequency, 10 sessions, each 15 min

SUMMARY:
The purpose of this study is to determine whether neurofeedback training can significantly reduce the symptoms of anorexia nervosa (AN) with focus on changes in personality and psychological well-being. The primary aims of this study include:

1. To examine whether AN patients are able to control their alpha-activity through neurofeedback.
2. To examine the effects of neurofeedback on symptomatology and personality variables in AN patients.
3. To examine the long-term effects of neurofeedback in the treatment of AN.

DETAILED DESCRIPTION:
The aim of the present study is to investigate the impact of EEG frequency band biofeedback (neurofeedback) training on EEG topography and symptomatology of patients suffering from anorexia nervosa (AN).

There is evidence that alpha-neurofeedback leads to an increase in positive therapy outcome in clinical populations by changing long-lasting EEG frequency patterns. The use of an EEG-guided relaxation paradigm has been shown to be associated with well-being and improvements in pathology of psychiatric patients.

In the present study the effects of alpha-training on EEG activity, mood, personality, well-being, blood parameters, and heart frequency will be evaluated in a sample of anorectic girls (12-18 years).

The subjects are trained with at least 10 sessions alpha-neurofeedback, in order to enhance individual alpha frequency, with spectral resting EEG, EKG, blood samples, ERP-measures and psychometric measures assessed before and after training. Neurofeedback is conducted over a period of five weeks, with each participant receiving two training sessions per-week. Neurofeedback is administered using USBAmp-EEG system.

For better surveillance of training effects there are two non-treatment control groups. A patient group receiving conventional therapy programme of the Psychosomatic Division of the Pediatric Department at the University Hospital Graz and a healthy control group.

A twelve-week follow-up study is carried out in order to document long-term effects of alpha-neurofeedback training in AN patients.

ELIGIBILITY:
Inclusion Criteria:

* anorexia nervosa diagnosed by ICD-10

Exclusion Criteria:

* epilepsy or other brain organic diseases

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
brain activity in the alpha band | 10 sessions neurofeedback
  measuring selected variables pre/posttraining and follow-up and on 10 points of measurement (10 sessions neurofeedback)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Lackner, Mag., Principal Investigator — Department of Psychology, Karl-Franzens-University Graz